CLINICAL TRIAL: NCT06796751
Title: PREcision Diagnostics in Rare genetIC Diseases and Tumors - Long Read Sequencing
Acronym: PREDICT-LRS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PREDICT-LRS; PNRR2022 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Whole Exome Sequencing; Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients with CNVs of unknown significance: The first subgroup of patients are those with SVs of unknown significance or uncertain disease mechanism.
  Interventions: Genetic: DNA/RNA sequencing and bioinformatic data analysis
- Patients with complex genomic rearrengements: Other complex rearrangements can be studied with LRS (i.e. ring chromosomes, isochromosome, chromosomal translocations, somatic SV found in tumors, etc.) to gain a better understanding of the molecular mechanisms of pathogenicity.
  Interventions: Genetic: DNA/RNA sequencing and bioinformatic data analysis
- Patients with a monoallelic variant in an AR gene: A third subgroup of patients eligible for the study are those with identified monoallelic alteration in autosomal recessive (AR) genes.
  Interventions: Genetic: DNA/RNA sequencing and bioinformatic data analysis
- Patients with negative results at WES analysis: Lastly, patients with a phenotype that is strongly suggestive for a genetic condition, in whom several analyses, including WES, retrieved negative results, could benefit from LRS.
  Interventions: Genetic: DNA/RNA sequencing and bioinformatic data analysis

INTERVENTIONS:
Genetic: DNA/RNA sequencing and bioinformatic data analysis — DNA will be extracted from peripheral blood or from somatic tissues. In some cases a skin biopsy will be performed to obtain fibroblasts for further analysis (DNA/RNA extraction and preparation of cell culture for high-throughput genomic and epigenomic technique (Hi-C).
  LRS will be performed on extracted DNA using Oxford Nanopore Technology by two different approaches:
  * Target, in samples with monoallelic alterations in genes related to autosomal recessive disease;
  * Genomic in other cases.
  Sequencing data will be analyzed through a dedicated bioinformatics pipeline, to reconstruct the tridimensional structure of chromatin and the regions

SUMMARY:
Using long-read sequencing (LRS) technology to achieve molecular diagnosis in patients with rare genetic diseases who have already been tested by state-of-the-art genetic analysis with ambiguous or negative results. This will lead to efficient and reliable identification and clinical interpretation of cryptic and complex structural genomic variants, which represent the central challenge for the coming decades in human genetics.

DETAILED DESCRIPTION:
The application of LRS to a diagnostic setting could have an impact on detection rate and diagnostic yield, leading to a better understanding of the etiology, prognosis and recurrence risk of rare genetic diseases (RGD), but also to a targeted treatment. One of the main benefits of LRS is the detection of balanced and unbalanced structural variants (SVs), including complex rearrangements, with high sensitivity and accuracy, through reliable alignment and precise breakpoint definition.

Among the main challenges of modern genetics, are identified 4 subgroups of patients that would benefit from the application of LRS to better characterize the genetic diagnosis and disease mechanisms.

* The first subgroup of patients are those with SVs of unknown significance or uncertain disease mechanism. In particular, clinical interpretation of duplications is challenging, due to the inability of Array Comparative Genomic Hybridization (aCGH) to detect whether they occur in tandem or are duplicated and inserted elsewhere in the genome, thus possibly disrupting genes involved in the duplication or altering their regulation.
* Other complex rearrangements can be studied with LRS to gain a better understanding of the molecular mechanisms of pathogenicity. A better definition of complex SVs, together with an accurate description of the phenotype, will allow the genotype-phenotype correlation to be determined.
* A third subgroup of patients eligible for the study are those with identified monoallelic alteration in autosomal recessive (AR) genes. The aim is to conduct a targeted analysis of the specific gene in order to look for a second mutation that wasn't detected by previous analysis (i.e. intronic variants, SVs, variants in difficult genomic regions).
* Lastly, patients with a phenotype that is strongly suggestive for a genetic condition, in whom several analyses, including Whole Exome-Sequencing (WES), retrieved negative results, could benefit from LRS. In this context, the aim is to apply a whole genome LRS approach to identify missed coding variants in difficult-to-sequence regions, variants in non-coding regions or SVs.

ELIGIBILITY:
Inclusion Criteria:

* patients/relatives of patients with Copy Number Variations (CNVs), previously detected by aCGH, with uncertain clinical significance;
* patients/relatives of patients with inconclusive WES and aCGH data (no pathogenic/likely pathogenic variant);
* patients/relatives of patients with a known single hit (a pathogenic or likely pathogenic variant) in an AR gene detected with WES or aCGH;
* patients/relatives of patients with a finding of complex structural variants whose molecular disease mechanism is to be elucidated.

Exclusion Criteria:

* none

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include:
  * patients previously in diagnostic routine, who have provided informed consent for storage and secondary use of their biological samples and for being recontacted; they will be informed about the current project and requested to provide a new specific informed consent;
  * patients' parents, when segregation analysis is required for diagnostic purpose; they will be informed about the current project and requested to provide a new specific informed consent;
  * age: from 0 years (newborns) with no upper age limit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The first aim of this study is to use LRS to reach a molecular diagnosis in patients with RGD that were already tested with state-of-the-art genetic analysis, with ambiguous or negative results. | 10 months
  In patients with RGD that were already tested with state-of-the-art genetic analysis, with ambiguous or negative results, will be use LRS to detect cryptic genomic variants that couldn't be detected with previous techniques. Clinical information of patients will be collected and integrated with genetic data.

SECONDARY OUTCOMES:
The secondary objective of this study is to analyze with a multi-omics approach, through the integration of other technologies supporting LRS (e.g. Hi-C, RNAseq), cases of particular complexity in which the molecular causative mechanism of the phenotype | 10 months
  Definition and precise characterization of structural variants and complex rearrangements with implication for their molecular diagnosis and clinical management.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Pippucci, Biologist, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No